CLINICAL TRIAL: NCT01602718
Title: Physical Activity and Functioning in Home Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Patricia Painter, Associate Research Faculty, University of Utah
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00053828
Record Dates: First submitted 2012-05-16; First posted 2012-05-21 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes
Keywords: physical activity; physical performance; ESRD; home dialysis
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity; Kidney Failure, Chronic | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Physical Function/Activity (No Intervention): cross-sectional comparison study of physical function/activity, frailty and inflammation measures in prevalent home Dx and prevalent in-center hemodialysis patients.
  Subjects: Forty-five prevalent home dialysis patients will be recruited and tested once for all outcome measures. Forty-five prevalent in-center hemodialysis patients will be identified from prevalent patients in the University of Utah in-center dialysis system who are matched for gender, age, comorbidities and time on dialysis as the home dialysis patients who have been tested. Consenting patients will be tested for all outcome measures once and compared to the home dialysis group.
- Incident Patients (No Intervention): Study 2: is a longitudinal cohort study of incident patients starting either home dialysis or in-center hemodialysis.
  Consenting patients will be tested upon initiation of dialysis therapy and every 6 months for 18 months to track physical functioning /activity, frailty and inflammation over time.
- Independent Home Exercise (Other): pilot study of independent home exercise training in home dialysis (PD only) patients. Consenting patients will be tested at baseline, then randomized into exercise training or usual care (no prescribed change in activity levels) and retested after 3 months.
  Interventions: Other: exercise training

INTERVENTIONS:
Other: exercise training — Pilot study of independent home exercise training (walking or cycling exercise plus low level resistance exercise) for 3 months. Patients will be given specific recommendations for type, frequency, duration and progression of their program and will be contacted weekly by study staff to assess progress and evaluation for any problems. This is a 3 month exercise training intervention in 15 subjects (and 15 no-exercise controls).
  Other Names: Independent Home Exercise Training
  Arms: Independent Home Exercise

SUMMARY:
This study will compare physical activity levels and physical functioning in patients treated with home dialysis vs. those treated with in-center dialysis. The investigators will first compare prevalent patients, and will also compare the two groups longitudinally in incident patients over the first 18 months of beginning the dialysis treatments. Patients will be tested for physical functioning using standard performance-based testing such as gait speed, chair stand, balance test, as well as self-reported limitations in activities of daily living. The investigators will monitor physical activity using step counters and activity questionnaires. Blood samples will be drawn at each testing time to measure inflammatory markers. A pilot study of home dialysis patients will be done to determine the effects of an independent home-based exercise program on physical functioning and inflammatory markers. For this pilot study, 30 patients will be randomized into exercise intervention and usual care with testing at baseline and again after 3 months of the intervention.

DETAILED DESCRIPTION:
Aim 1: To determine levels of physical functioning, physical activity, incidence of frailty and inflammation status in prevalent home dialysis patients in the University of Utah Home Dialysis program and compare them to in-center hemodialysis patients who are matched for age, gender, comorbidities and dialysis vintage. Hypothesis 1: Patients on home therapies will have higher physical functioning, be more active and fewer will be frail compared to matched patients treated with in-center hemodialysis.

Aim 2: To determine the patterns of change in physical functioning and physical activity over the first 18 months of initiating dialysis therapy. Hypothesis 2: Physical functioning and physical activity will be maintained in patients initiating home dialysis therapy, whereas, those initiating in-center dialysis will deteriorate in physical functioning and physical activity.

Aim 3: To determine the effects of counseling and encouragement of physical activity in prevalent home dialysis patients on physical functioning, physical activity. Hypothesis 3: Compared to usual care, patients who are counseled and encouraged to participate in independent home walking exercise will improve physical functioning and health-related quality of life.

Aim 4: To determine the association of inflammation with physical functioning in home dialysis patients and with changes in physical activity. Hypothesis 4: Lower physical functioning is associated with inflammation and increased physical activity will improve physical functioning and reduce the associated inflammation.

ELIGIBILITY:
Inclusion Criteria:

* on dialysis for 3 months (for prospective study and for pilot intervention)
* 18 years of age
* ambulatory
* no progressive neuromuscular disease
* no orthopedic or rheumatologic problems that would be exacerbated by physical function testing
* English speaking
* able to understand and provide consent for participation

Exclusion Criteria:

* progressive neuromuscular disease that may result in limitations
* orthopedic or rheumatologic disease that may be exacerbated by physical function testing
* physical functioning
* unstable angina or angina upon exertion
* terminal illness with life expectancy less than 12 months
* MI or CABG within the last year
* NYHA Class III or IV CHF

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
change in short physical performance battery | baseline, 3 months, 6 months 12 mo, 18 mo

SECONDARY OUTCOMES:
change in inflammation | baseline, 6 mo, 12 mo, 18 mo

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Painter, Principal Investigator — U of U PHYSICAL THERAPY - COH

REFERENCES:
- [Background] Painter P, Carlson L, Carey S, Paul SM, Myll J. Physical functioning and health-related quality-of-life changes with exercise training in hemodialysis patients. Am J Kidney Dis. 2000 Mar;35(3):482-92. doi: 10.1016/s0272-6386(00)70202-2. PMID 10692275
- [Background] Lo CY, Li L, Lo WK, Chan ML, So E, Tang S, Yuen MC, Cheng IK, Chan TM. Benefits of exercise training in patients on continuous ambulatory peritoneal dialysis. Am J Kidney Dis. 1998 Dec;32(6):1011-8. doi: 10.1016/s0272-6386(98)70076-9. PMID 9856517
- [Background] Painter P, Messer-Rehak D, Hanson P, Zimmerman SW, Glass NR. Exercise capacity in hemodialysis, CAPD, and renal transplant patients. Nephron. 1986;42(1):47-51. doi: 10.1159/000183632. PMID 3510400
- [Background] Cheema BS, Singh MA. Exercise training in patients receiving maintenance hemodialysis: a systematic review of clinical trials. Am J Nephrol. 2005 Jul-Aug;25(4):352-64. doi: 10.1159/000087184. Epub 2005 Jul 22. PMID 16088076